CLINICAL TRIAL: NCT06787742
Title: Assessment of the Number of Missing Tooth Surfaces and a New Bioceramic Material on the Outcomes of Vital Pulp Therapy: A Randomized Clinical Study
Brief Title: Assessment of the Number of Missing Tooth Surfaces and the Molecular Findings on the Outcomes of Vital Pulp Therapy Using Two Calcium Silicate Materials
Acronym: VPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (528/2022)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Vital Pulp Therapies; Tooth Defect
Keywords: Biomarkers; Calcium silicate cements; Full pulpotomy; Irreversible pulpitis; Mature teeth
MeSH Terms: interventions — Hemostasis

STUDY DESIGN:
Intervention Model Description: A comparative, randomized, prospective clinical study was utilized for the investigation of the outcome of pulpotomy in the treatment of adult permanent mandibular molar teeth with symptomatic irreversible pulpitis in class I and class II cavity defects using two types of hydraulic calcium silicate cement (MTA+) and (Well-root PT)
Who Masked: Participant, Investigator
Masking Description: did not inform the patients which type of material was used, All laboratory procedures were performed by a single, experienced individual specializing in biochemical assays, without informing the biochemist of any outcome data of pulpotomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A. Number of tooth surfaces defects: • Class I cavity defect. • Class II cavity defect. (Active Comparator): The selected patients were divided into two groups according to the number of tooth surfaces defects (n=30) (30 with class I and 30 with class II cavity defects)
  Interventions: Procedure: full pulpotomy
- pulpotomy dressing materials: • MTA+ (Cerkamed, Poland). • Well-Root (Vericom, Korea). (Active Comparator): Each group was randomly further subdivided using Microsoft Excel into two subgroups according to the dressing materials, without informing the patients which type of material was used (n=15).
  Interventions: Procedure: full pulpotomy

INTERVENTIONS:
Procedure: full pulpotomy — access to dental pulp chamber under aseptic condition, collect blood sample using a micropipette for ELIZA test, stop bleeding using sodium hypochlorite 2.5%, pulpotomy dressing material over pulp stump and final restoration with resign modified glass ionomer and composite resign
  Other Names: collecting pulpal blood samples; Hemostasis; pulpotomy dressing materials; final restoration

SUMMARY:
The present study aimed to evaluate and compare the clinical and radiographic outcomes of full pulpotomy in mandibular molar teeth with symptomatic irreversible pulpitis according to:

A. Number of tooth surfaces defects:

* Class I cavity defect.
* Class II cavity defect.

B. Using two types of pulpotomy dressing materials:

* MTA+ (Cerkamed, Stalowa, Poland).
* Well-Root PT (Vericom, Gangwon-Do, Korea). And.,

To correlate this outcome to the quantification of two biomolecules:

* Tumor necrosis factor-alpha (TNF-⍺).
* Matrix metalloproteinases-9 (MMP-9).

Based on the results of the present study, it was concluded that:

1. Full pulpotomy using calcium silicate cements (CSCs) is considered a conservative, economical, and simple treatment option with a favorable prognosis for teeth with symptomatic irreversible pulpitis.
2. Class I and class II cavity defects do not adversely affect pulpotomy prognosis taking into consideration good aseptic condition, magnification, and proper seal of filling materials.
3. Although MTA+ and Well-Root PT yielded similar outcomes for pulpotomy in terms of success rates. Well-root PT is easier to handle compared to MTA+ and doesn't have a discoloration effect which is considered one of the drawbacks associated with MTA+.
4. Neither the preoperative pain nor the intraoperative bleeding time within 10 minutes influenced the pulpotomy outcome.
5. The concentration of TNF-α and MMP-9 biomarkers directly impact the outcome of pulpotomy.

DETAILED DESCRIPTION:
The current study addresses an important gap in research, as the impact of cavity configuration on the outcomes of full pulpotomy has not been well explored. Comparing Class I and Class II cavity defects in this context can provide valuable insights, especially given the differences in structural integrity, bacterial infiltration risks, and restorative challenges associated with these defects.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular molar teeth with signs and symptoms of symptomatic irreversible pulpitis without radiographic evidence of apical periodontitis.
* Age range of 21-45 years old.
* Males or females.
* No disabilities.
* Class I and/or class II cavity defects.
* Teeth reveal positive response to cold tests.

Exclusion Criteria:

* Presence of open apices.
* Non-restorable teeth.
* Teeth in which the pulpal bleeding time is more than 10 minutes.
* Presence of large carious lesions approaching the root.
* Presence of calcification or resorption.
* Periodontally affected teeth.
* Patients who are taking antibiotics within one week before treatment.
* Patients consumed taking analgesics within 24 hours before treatment.
* Systemically compromised patients.
* Pregnant females.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
success/failure | Patients were scheduled for follow-up appointments (one week, 3, 6, and 12 months)
  Treatment was considered successful (healed) according to Zanini et al. (2016) based on the following criteria:
  (Clinically) absence of signs and symptoms of pulpal pathosis, no history of spontaneous pain or discomfort on chewing, no tenderness to percussion/palpation, no soft tissue swelling, fistula, or abnormal mobility. (Radiographically) absence of periapical rarefaction (normal width of periodontal ligament space and normal appearance of the lamina dura), internal or external resorption, and absence of root canal calcification
Pain assessment | every 24 hours in the evening for 7 days
  Pre-treatment, the patients were instructed on how to fill out a visual analog scale VAS to determine their pain score. Postoperative pain was recorded by the patient every 24 hours in the evening for 7 days. The VAS included scores from 0 to 10, which were further categorized as no pain (0), mild (1-3), moderate (4-6), severe (7-9), or severe intolerable (10).

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Mukhtar Fayyad, Professor of endodontics, Study Chair — Suez Canal University
Locations (1):
- Faculty of Dentistry, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided